CLINICAL TRIAL: NCT03383666
Title: A Prospective, Multi-center, Single Arm Study to Evaluate the Safety and Effectiveness of the PulseRider® Aneurysm Neck Reconstruction Device Used in Conjunction With Endovascular Coil Embolization in the Treatment of Wide-Neck Bifurcation Intracranial Aneurysm
Brief Title: A Study Evaluating the Safety and Effectiveness of the PulseRider® Aneurysm Neck Reconstruction Device Used in Conjunction With Endovascular Coil Embolization in the Treatment of Wide-Neck Bifurcation Intracranial Aneurysm
Acronym: NAPA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No safety issues; change in innovation strategy
Sponsor: Pulsar Vascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSC_2017-01
Record Dates: First submitted 2017-12-12; First posted 2017-12-26 (Actual); Results first posted 2022-04-14 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Unruptured Wide-neck Intracranial Aneurysms
Keywords: Unruptured; intracranial aneurysms; Endovascular
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Group (Experimental): PulseRider® Aneurysm Neck Reconstruction in conjunction with coil embolization for unruptured wide-neck intracranial aneurysms.
  Interventions: Device: PulseRider® Aneurysm Neck Reconstruction Device

INTERVENTIONS:
Device: PulseRider® Aneurysm Neck Reconstruction Device — Neck Reconstruction Device

SUMMARY:
This is a prospective, multi-center, non-randomized clinical evaluation utilizing the PulseRider® Aneurysm Neck Reconstruction Device.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and effectiveness of the PulseRider® Aneurysm Neck Reconstruction Device in conjunction with coil embolization in the endovascular treatment of unruptured wide-neck intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with wide neck intracranial aneurysm located at a bifurcation
2. The subject is between 18 and 80 years of age the time of consent
3. Informed consent is obtained and the subject signs the IRB approved consent prior to beginning any study procedures
4. In the opinion of the treating physician, placement of the PulseRider® device is technically feasible and clinically indicated

Exclusion Criteria:

1. Unstable neurological deficit (condition worsening within the last 90 days)
2. Subarachnoid Hemorrhage (SAH) within the last 60 days
3. Irreversible bleeding disorder
4. Patient has another intracranial aneurysm that in the Investigator's opinion, may require treatment within the 1 year follow up period
5. A history of contrast allergy that cannot be medically controlled
6. Known allergy to nickel
7. Relative contraindication to angiography
8. Woman of child-bearing potential who cannot provide a negative pregnancy test
9. Current involvement in a study for another investigational product
10. Patient and / or family considering a move from this geographical location at the time of consent
11. Categorized as a vulnerable population and require special treatment with respect to safeguards of well-being (e.g. cognitively impaired, veteran, prisoner, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mount Sinai Hospital, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- PulseRider Aneurysm Neck Reconstruction Device: Participants with wide-neck bifurcation intracranial aneurysms were implanted with PulseRider device.
Period: Overall Study
Arm/Group | PulseRider Aneurysm Neck Reconstruction Device
Started | 21
Implanted With Pulse Rider | 18
Attempted But Unsuccessful Implantation | 3
Completed | 17
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: The modified intent to treat (mITT) analysis set is defined as all enrolled participants in whom treatment with the PulseRider device was attempted as defined by advancement of any portion of the PulseRider device outside of the distal end of the microcatheter inside the participant.
Arm/Group | PulseRider Aneurysm Neck Reconstruction Device
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Aneurysm Occlusion Without Significant Parent Artery Stenosis or Prior Retreatment Through 1 Year Post-Procedure
Description: Number of participants with complete aneurysm occlusion (Raymond I: complete occlusion) without significant parent artery stenosis (greater than [>] 50 percent [%] stenosis) or prior retreatment through 1-year post procedure were reported.
Time Frame: Up to 1 year post procedure
Population: The Per Protocol (PP) analysis set is defined as all participants successfully implanted with the PulseRider device with no major protocol deviations. Here, N (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PulseRider Aneurysm Neck Reconstruction Device
Number analyzed (Participants) | 13
Participants | 10

2. Primary Outcome: Percentage of Participants With Occurrence of Neurological Death or Major Ipsilateral Stroke in Downstream Territory up to 1 Year Post-procedure Per Clinical Events Committee (CEC)
Description: Percentage of participants with occurrence of neurological death or major ipsilateral stroke in downstream territory up to 1 year post-procedure per CEC were reported. Major stroke is defined as stroke with symptoms persisting for more than 24 hours and a sudden increase in the National Institutes of Health Stroke Scale (NIHSS) of the subject by greater than or equal to (>=) 4. Major ipsilateral stroke is major stroke in downstream territory.
Time Frame: Up to 1 year post procedure
Population: The modified intent to treat (mITT) analysis set is defined as all enrolled participants in whom treatment with the PulseRider device was attempted as defined by advancement of any portion of the PulseRider device outside of the distal end of the microcatheter inside the participant. Here, N (number of participants analyzed) defined as participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | PulseRider Aneurysm Neck Reconstruction Device
Number analyzed (Participants) | 17
Percentage of Participants
  Major Ipsilateral Stroke in Downstream Territory | 0
  Neurological Death | 0

3. Secondary Outcome: Number of Participants With Technical Success of Successful Implantation of the PulseRider Device
Description: Technical success was defined as successful implantation of the PulseRider device- the ability to access the target aneurysm, deploy the device at the aneurysm neck, and detach device successfully. Number of participants with technical success were reported.
Time Frame: Up to 1 year
Population: The mITT analysis set is defined as all enrolled participants in whom treatment with the PulseRider device was attempted as defined by advancement of any portion of the PulseRider device outside of the distal end of the microcatheter inside the participant.
Measure: Count of Participants; unit: Participants
Arm/Group | PulseRider Aneurysm Neck Reconstruction Device
Number analyzed (Participants) | 21
Participants | 18

4. Secondary Outcome: Number of Participants With Target Aneurysms Retreatment
Description: Number of participants with target aneurysms retreatment were reported.
Time Frame: Up to 1 year
Population: The PP analysis set is defined as all participants successfully implanted with the PulseRider device with no major protocol deviations from the eligibility criteria or dual antiplatelet medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PulseRider Aneurysm Neck Reconstruction Device
Number analyzed (Participants) | 17
Participants | 0

5. Secondary Outcome: Number of Participants With Significant Stenosis (>50%) at Implant Site
Description: Number of participants with significant stenosis (>50%) at implant site were reported.
Time Frame: Up to 1 year
Population: The PP analysis set is defined as all participants successfully implanted with the PulseRider device with no major protocol deviations. Here, N (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PulseRider Aneurysm Neck Reconstruction Device
Number analyzed (Participants) | 13
Participants | 0

6. Secondary Outcome: Number of Participants With Adequate Aneurysm Occlusion
Description: Number of participants with adequate aneurysm occlusion were reported.
Time Frame: 1 year
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | PulseRider Aneurysm Neck Reconstruction Device
Number analyzed (Participants) | 13
Participants | 13

7. Secondary Outcome: Number of Participants With Modified Rankin Scale (mRS) 0-2
Description: Number of participants with modified rankin scale (mRS) 0-2 were reported. The mRS is a scale commonly used to measure the degree of disability or dependence in the daily activities in patients following stroke or other neurologic event and is conducted by qualified personnel. It is a scale with six categories ranging from no symptoms to severe disability and death.
Time Frame: 1 year
Population: The PP analysis set is defined as all participants successfully implanted with the PulseRider device with no major protocol deviations from the eligibility criteria or dual antiplatelet medication. Here, N (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PulseRider Aneurysm Neck Reconstruction Device
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Time Frame: From enrollment up to 1 year post procedure.
Description: Modified intent to treat (mITT) analysis set: all enrolled Participants in whom treatment with PulseRider device was attempted. Adverse event data was adjudicated by independent Clinical Events Committee (CEC).
Arm/Group | PulseRider Aneurysm Neck Reconstruction Device
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PulseRider Aneurysm Neck Reconstruction Device (N=21)
Pneumonia (Infections and infestations) | 2
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PulseRider Aneurysm Neck Reconstruction Device (N=21)
Migraine (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1
Diplopia (Eye disorders) | 2
Eye haemorrhage (Eye disorders) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Confusional state (Psychiatric disorders) | 1
Hallucination, visual (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Asthenia (General disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
Only 1-year endpoint analyses were performed due to early termination of study enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT03383666/Prot_SAP_004.pdf